CLINICAL TRIAL: NCT02896413
Title: The Effects of Perioperative Dexmedetomidine Administration on Immune Suppression and Outcomes in Patients With Uterine Cancer Undergoing Radical Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 4-2015-0453
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Uterine Cancer
MeSH Terms: conditions — Uterine Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine Group (Experimental): dexmedetomidine infusion (0.4 mcg/kg/h) from immediately after anesthetic induction to 24 h after surgery
  Interventions: Drug: Dexmedetomidine group
- Control Group (Placebo Comparator): 0.9% saline infusion
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Dexmedetomidine group — dexmedetomidine infusion (0.4 mcg/kg/h) from immediately after anesthetic induction to 24 h after surgery
  Arms: Dexmedetomidine Group
Drug: Control group — 0.9% saline infusion
  Arms: Control Group

SUMMARY:
Surgical stress and anesthesia may cause immunosuppression in immunocompromised cancer patients. The natural killer (NK) cell is a critical part of anti-tumor immunity. Dexmedetomidine has sympatholytic effect and preserves NK cell function. This study investigate the effect of dexmedetomidine on immune suppression and postoperative outcomes in patients undergoing uterine cancer resection.

ELIGIBILITY:
Inclusion Criteria:

* patient between 20 and 70 of age with ASA physical status Ⅰ-Ⅲ
* patient scheduled for uterine cancer surgery

Exclusion Criteria:

* ASA physical status Ⅳ
* severe hepatorenal disease
* infection
* metastasis to other organ
* problem with communication

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
natural killer cell cytotoxicity | 1 minute before surgery
  Natural killer cell cytotoxicity is measured with NK Vue Kit™(ATGen, Gyeonggi-do, Korea).
natural killer cell cytotoxicity | postoperative day 1
  Natural killer cell cytotoxicity is measured with NK Vue Kit™(ATGen, Gyeonggi-do, Korea).
natural killer cell cytotoxicity | postoperative day 3
  Natural killer cell cytotoxicity is measured with NK Vue Kit™(ATGen, Gyeonggi-do, Korea).
natural killer cell cytotoxicity | postoperative day 5
  Natural killer cell cytotoxicity is measured with NK Vue Kit™(ATGen, Gyeonggi-do, Korea).

SECONDARY OUTCOMES:
inflammatory response | 1 minute before surgery
  inflammatory response is assessed by measuring levels of proinflammatory cytokines.
inflammatory response | postoperative day 1
  inflammatory response is assessed by measuring levels of proinflammatory cytokines.
inflammatory response | postoperative day 3
  inflammatory response is assessed by measuring levels of proinflammatory cytokines.
inflammatory response | postoperative day 5
  inflammatory response is assessed by measuring levels of proinflammatory cytokines.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No